CLINICAL TRIAL: NCT03693144
Title: Location Initiated Individualized Texts for African American Adolescent Health
Brief Title: Improving Nutritional Choices in Adolescents
Acronym: LIITA3H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Susan J Woolford, MD, MPH, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HUM00083980; 1R21HD093835-01 (NIH)
Record Dates: First submitted 2018-09-28; First posted 2018-10-02 (Actual); Results first posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-09

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group 1 Full LIITA3H App (Experimental): Participants were given the LIITA3H app, which is a combination product consisting of 3 main features that tracked their visits to fast food restaurants (using the ELI feature), sent tailored text messages to prompt healthy choices when they were in a fast food restaurant (using the POP feature), and allowed them to submit pictures of their food (using the SNAP feature).
  Interventions: Other: Full LIITA3H App
- Control Group 2 Partial LIITA3H App (Active Comparator): Participants were given the LIITA3H app that tracked their visits to fast food restaurants (using the ELI feature) and they submitted pictures of their food (using the SNAP feature). However, they did not receive tailored text messages.
  Interventions: Other: Partial LIITA3H App
- Control Group 3 LIITA3H Location only (Other): Participants were given the LIITA3H app that tracked their visits to fast food restaurants (using the ELI feature) but they did not receive tailored messages or submit pictures of their food.
  Interventions: Other: LIITA3H Location only

INTERVENTIONS:
Other: Full LIITA3H App — This is the full version of the LIITA3H mobile app that will use the Enhanced Location Identification (ELI) technology to identify when a user is in an eating venue and then deliver culturally and individually tailored point of purchase prompts (POP) to encourage healthy choices and will allow participants to take pictures of the food they purchase using the Self-report of Nutrients with Annotated Photos (SNAP) function.
  Arms: Intervention Group 1 Full LIITA3H App
Other: Partial LIITA3H App — This is a version of the LIITA3H mobile app that will track participants' location and allow them to submit photos of their food.
  Arms: Control Group 2 Partial LIITA3H App
Other: LIITA3H Location only — This is a version of the LIITA3H mobile app that will only track participants' location.
  Arms: Control Group 3 LIITA3H Location only

SUMMARY:
The goal of this project is to test whether the mobile application helps Black adolescents make healthy food choices at the point of purchase.

DETAILED DESCRIPTION:
The epidemic of excess weight in childhood is impacted by exposure to, and consumption of, fast food and calorie dense foods prepared outside of the home. Black youth are more likely than their peers to live in communities with a high density of fast food restaurants. There is a need for interventions to help adolescents make healthy choices in these obesogenic environments.

Previous research revealed that adolescents welcomed health-related text messages (based on Self Determination Theory and Motivational Interviewing) if they viewed them as personally relevant and if they were received at times when they faced dietary choices. Based on these findings, the following is hypothesized: that delivering messages (tailored to users' preferences and values) at a time and place when they are making a dietary choice (e.g., in a restaurant) will positively influence their choices.

Thus, the Location Initiated Individualized Texts for African American Adolescent Health (LIITA3H) mobile application was developed. This app identifies when users were in a restaurant, automatically sends culturally relevant messages (based on focus group input from the target population) tailored to user preferences and the menu options at their location with the aim of prompting users to make a healthy choice, and allows users to submit an annotated photo response about their food choice.

For this R21 project the following will be achieved: 1) the LIITA3H app will be enhanced by incorporating user input regarding its design and by allowing greater automation in the identification of eating venues, and 2) the impact of the app on the number of visits by users to restaurants, and on the number of calories users consume from these venues will be tested. This will provide data regarding effect size and will form the foundation for a large randomized trial in a larger population and including a greater range of eating venues. A better understanding of how 'just in time" personalized cues to action, made possible by new location-based technology, might alter behavior among a high risk population, will help future efforts to address obesity and other illnesses impacted by lifestyle choices.

As of 2020, due to the influence of the public health emergency, lockdowns prevented any participants from engaging in going to restaurants as they previously would have. Due to the trial beginning in November 2019, no six month app based data was acquired before the lockdown, and research limitations were imposed. When behavioral research of this type was allowed to resume, months later, a very limited time remained before the funded study would have to end. Thus, certain aspects of the protocol and intervention were modified. To be pragmatic under these constrained circumstances, for new participants, the intervention was shortened from 6 months to 1 month. As behavioral change takes longer to be achieved, the 1 month abbreviated trial focused on exploring the functionality of the app to lay the groundwork for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Self identification as African American
* BMI at or above 85th percentile
* Eat at fast food restaurants at least 3 times per week at baseline

Exclusion Criteria:

-

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Woolford, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group 1 Full LIITA3H App: Participants were given the LIITA3H app, which is a combination product consisting of 3 main features that: tracks their visits to fast food restaurants (using the ELI feature), sends tailored text messages to prompt healthy choices when they are in a fast food restaurant (using the POP feature), and allows them to submit pictures of their food (using the SNAP feature).
  Full LIITA3H App: This is the full version of the LIITA3H mobile app that used the Enhanced Location Identification (ELI) technology to identify when a user is in an eating venue and then deliver culturally and individually tailored point of purchase prompts (POP) to encourage healthy choices and allows participants to take pictures of the food they purchase using the Self-report of Nutrients with Annotated Photos (SNAP) function.
- Control Group 2 Partial LIITA3H App: Participants were given the LIITA3H app that tracks their visits to fast food restaurants (using the ELI feature) and they could submit pictures of their food (using the SNAP feature). However, they did not receive tailored text messages.
  Partial LIITA3H App: This is a version of the LIITA3H mobile app that tracks participants' location and allows them to submit photos of their food.
- Control Group 3 LIITA3H Location Only: Participants were given the LIITA3H app that tracks their visits to fast food restaurants (using the ELI feature) but they did not receive tailored messages or submit pictures of their food.
  LIITA3H Location only: This is a version of the LIITA3H mobile app that only tracks participants' location.
Period: Overall Study
Arm/Group | Intervention Group 1 Full LIITA3H App | Control Group 2 Partial LIITA3H App | Control Group 3 LIITA3H Location Only
Started | 7 | 7 | 5
Completed (Completion = maintaining the app on their phone, or participating in an end-of-study interview, but as COVID shut down Fast Food Restaurants approximately four months after the first enrollment, no six-month data could be gathered from the app.) | 7 | 5 | 4
Not Completed | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group 1 Full LIITA3H App | Control Group 2 Partial LIITA3H App | Control Group 3 LIITA3H Location Only | Total
Number analyzed (Participants) | 7 | 7 | 5 | 19
Age, Continuous [Mean (Full Range); unit: years] | 15 [13 to 17] | 14 [13 to 17] | 15 [13 to 17] | 15 [13 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 2 | 13
  Male | 1 | 2 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 7 | 5 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 7 | 5 | 19
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 5 | 19

OUTCOME MEASURES:

1. Primary Outcome: Visits to Fast Food Restaurants
Description: Change in number of weekly visits to Fast Food Restaurants
Time Frame: Over 6 months
Population: Due to COVID changes forcing closure of Fast Food Restaurants and changes in restaurant indoor dining policies; along with changes in behavior associated with COVID-related lockdowns, no six month data for this outcome was acquired.
Arm/Group | Intervention Group 1 Full LIITA3H App | Control Group 2 Partial LIITA3H App | Control Group 3 LIITA3H Location Only
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Calories Purchased From Fast Food Restaurants
Description: Change in number of calories purchased per week at Fast Food Restaurants
Time Frame: After 6 months of app use
Population: Due to COVID changes forcing closure of Fast Food Restaurants and changes in restaurant indoor dining policies; along with changes in behavior associated with COVID-related lockdowns, no six month data for this outcome could be acquired.
Arm/Group | Intervention Group 1 Full LIITA3H App | Control Group 2 Partial LIITA3H App | Control Group 3 LIITA3H Location Only
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Percentage of Times App Identifies Presence in Fast Food Restaurant (FFR)
Description: Percentage of times the app correctly identifies that a participant is in a registered Fast Food Restaurant.
Time Frame: Over 6 months
Population: This was not analyzable due to problems with the technology employed. During the COVID truncated implementation of this trial, the means to allow participants to confirm or deny that they were in a Fast Food Restaurant when the app signaled that they were was not incorporated into the app appropriately. Comparably, the ability for them to tell us that they were in a Fast Food Restaurant but that the app failed to identify that location as a FFR was not incorporated into the app appropriately.
Arm/Group | Intervention Group 1 Full LIITA3H App | Control Group 2 Partial LIITA3H App | Control Group 3 LIITA3H Location Only
Number analyzed (Participants) | 0 | 0 | 0

4. Primary Outcome: Percentage of Times App Delivers Appropriate Tailored Message
Description: Percentage of times the app delivers a tailored message for a menu item at the Fast Food Restaurant in which the participant is located. (number of times a tailored message is delivered divided by the number of times the app identified that the user was in a Fast Food Restaurant x 100).
Time Frame: over 1 month
Population: The population consisted of participants in the intervention arm
Measure: Number; unit: percentage of times
Arm/Group | Intervention Group 1 Full LIITA3H App
Number analyzed (Participants) | 7
percentage of times | 100

5. Secondary Outcome: Participants' Perception of the Experience of Using the App
Description: Participants' perception of the acceptability of the app's content and design via qualitative assessment. While the original intent for this outcome measure was to assess perceptions after 6 months of app use, because of the constraints of COVID, these interviews were primarily performed after a single month in the study.
Time Frame: At the completion of at least 1 month in the study
Population: Participants who completed the study final assessment interview.
Measure: Count of Participants; unit: Participants
Groups:
- Control Group 2 LIITA3H Location Only: Participants were given the LIITA3H app that tracks their visits to fast food restaurants (using the ELI feature) but they did not receive tailored messages or submit pictures of their food.
  LIITA3H Location only: This is a version of the LIITA3H mobile app that only tracks participants' location.
Arm/Group | Intervention Group 1 Full LIITA3H App | Control Group 2 Partial LIITA3H App | Control Group 2 LIITA3H Location Only
Number analyzed (Participants) | 5 | 3 | 2
Participants
  Enjoyed Messages | 4 | NA — Control Groups did not receive messages, thus they were not asked this question. | NA — Control Groups did not receive messages, thus they were not asked this question.
  Possible Desire to Continue App Use | 4 | NA — Control Groups did not receive messages, thus they were not asked this question. | NA — Control Groups did not receive messages, thus they were not asked this question.
  Experienced at Least One Difficulty with App Functioning | 5 | 2 | 0

ADVERSE EVENTS:
Time Frame: From initial enrollment to last interview; due to COVID -required interruption in research the longest interval between these events was 18 months.
Arm/Group | Intervention Group 1 Full LIITA3H App | Control Group 2 Partial LIITA3H App | Control Group 3 LIITA3H Location Only
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT03693144/Prot_SAP_000.pdf